CLINICAL TRIAL: NCT04899258
Title: Effect of Myopic Femtosecond Laser Asssisted-LASIK on Anaterior Chamber Flare Values and Corneal Endothelial Cells
Brief Title: Evaluation of the Effect of Myopic Femtosecond Laser Assisted-LASIK on Anterior Chamber Flare Values and Corneal Endothelial Cells: A Prospective Before-and-After Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Kemal Turgay Ozbilen, M.D. Academics, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06.12.2019/20/1495
Record Dates: First submitted 2021-05-10; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Cornea; Refractive Surgery; Anterior Chamber Inflammation
Keywords: Excimer laser Corneal Endothelium; Laser in situ keratomileusis (LASIK);; femtosecond assisted-LASIK; Anterior chamber flare; Endothelial cell densit; Corneal Endothelium
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: prospective, before-after study
Masking Description: Patients name and identifiers were masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-surgery and post-surgery (Other): femtosecond assisted LASIK
  Interventions: Procedure: Femtosecond laser assisted LASIK

INTERVENTIONS:
Procedure: Femtosecond laser assisted LASIK — Refractive surgery

SUMMARY:
This study aimed to investigate whether femtosecond laser-assisted LASIK (FS-LASIK) surgery causes inflammation in the anterior chamber and to analyze its effect on endothelial cells.

DETAILED DESCRIPTION:
Since FS-LASIK surgery is applied using both an FS laser and an excimer laser, we aimed to determine the direct and indirect effects of these applications on the corneal endothelium, the intensity of the inflammation, and the blood-aqueous barrier in the anterior chamber. To the best of our knowledge, the effects of FS-LASIK on anterior chamber inflammation have not been previously investigated. Therefore, we evaluated these effects using objective measurement methods, such as specular microscopy and laser flare photometry.

ELIGIBILITY:
Inclusion Criteria:

* The patients who performed Femtosecond laser assisted LASIK for myopia or myopic astigmatism.
* Uncomplicated surgery

Exclusion Criteria:

* Complicated surgery,
* Hyperopic or hyperopic astigmatism
* Lack of follow-up measurements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change of Flare Values | The change of flare values on first day, seventh day, 1. month and 3. months according to preoperative values
  To measure anterior chamber inflammation objectively, Flare values were measured by the laser flare-photometry

SECONDARY OUTCOMES:
Change of Corneal endothelium features-1 | the changes of the parameters of preoperative and 3. months' values
  Endothelial cell density (ECD),(The parameter was measured by specular microscopy)

OTHER OUTCOMES:
Change of Corneal endothelium features-2 | the changes of the parameters of preoperative and 3. months' values
  Coefficient of Varience (CV) in cell size, (The parameter was measured by specular microscopy)
Change of Corneal endothelium features-3 | the changes of the parameters of preoperative and 3. months' values
  Hexagonality percent of the cell shape. (The parameter was measured by specular microscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Turgay Ozbilen, M.D., Principal Investigator — Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozbilen KT, Altinkurt E, Ceylan NA, Bilgin GS, Gozum N. Effect of Myopic Femtosecond Laser-Assisted LASIK on Anterior Chamber Inflammation (Flare Values) and Corneal Endothelium: A Prospective before and after Study. J Ophthalmol. 2021 Nov 26;2021:2395028. doi: 10.1155/2021/2395028. eCollection 2021. PMID 34868671